CLINICAL TRIAL: NCT02543567
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate A Range of Dose Levels of a Heterologous Prime-Boost Regimen of Ad26.ZEBOV and MVA-BN®-Filo in Healthy Adult Subjects
Brief Title: A Study to Evaluate A Range of Dose Levels of Ad26.ZEBOV and MVA-BN-Filo in Healthy Adult Participants
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Vaccines & Prevention B.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CR107861; VAC52150EBL3002 (Other: Janssen Vaccines & Prevention B.V.)
Record Dates: First submitted 2015-09-04; First posted 2015-09-07 (Estimated); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Healthy
Keywords: Ebola viruses; Ebola virus disease (EVD); Filoviruses; Monovalent vaccine; Safety; Immunogenicity; Ebola vaccine; Human adenovirus serotype 26 (Ad26) expressing the Ebola virus Mayinga variant glycoprotein (Ad26.ZEBOV); Modified Vaccinia Virus Ankara - Bavarian Nordic Filo-vector (MVA-BN Filo); Healthy participants
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1 (Experimental): Ad26.ZEBOV 5*10^10 viral particles (vp) single dose intramuscular (IM) injection on Day 1; MVA-BN-Filo 1*10^8 Infectious Unit [Inf. U.] single dose IM injection on Day 57
  Interventions: Biological: Ad26.ZEBOV 5*10^10 viral particles (vp); Biological: MVA-BN-Filo 1*10^8 Infectious Unit [Inf. U.]
- Group 2 (Experimental): Ad26.ZEBOV 2*10^10 vp single dose intramuscular (IM) injection on Day 1; MVA-BN-Filo 5*10^7 Inf. U single dose IM injection on Day 57
  Interventions: Biological: Ad26.ZEBOV 2*10^10 (vp); Biological: MVA-BN-Filo 5*10^7 Inf. U.
- Group 3 (Experimental): Ad26.ZEBOV 0.8*10^10 vp single dose intramuscular (IM) injection on Day 1; MVA-BN-Filo 5*10^7 Inf. U. single dose IM injection on Day 57
  Interventions: Biological: Ad26.ZEBOV 0.8*10^10 (vp); Biological: MVA-BN-Filo 5*10^7 Inf. U.
- Group 4 (Experimental): Participants will receive intramuscular (IM) injection of Placebo (0.9% saline) once on Day 1 and Day 57
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Ad26.ZEBOV 5*10^10 viral particles (vp) — Ad26.ZEBOV, live, replication incompetent vaccine, sterile suspension for intramuscular (IM) injection of 5*10^10 viral particles on Day 1
  Arms: Group 1
Biological: Ad26.ZEBOV 2*10^10 (vp) — Ad26.ZEBOV, live, replication incompetent vaccine, sterile suspension for intramuscular (IM) injection of 2*10^10 viral particles on Day 1
  Arms: Group 2
Biological: Ad26.ZEBOV 0.8*10^10 (vp) — Ad26.ZEBOV, live, replication incompetent vaccine, sterile suspension for intramuscular (IM) injection of 0.8*10^10 viral particles on Day 1
  Arms: Group 3
Biological: MVA-BN-Filo 1*10^8 Infectious Unit [Inf. U.] — MVA-BN-Filo- live replication incompetent vaccine, IM injection of 1*10^8 Infectious Unit [Inf. U.] once on Day 57
  Arms: Group 1
Biological: MVA-BN-Filo 5*10^7 Inf. U. — MVA-BN-Filo- live replication incompetent vaccine, IM injection of 5*10^7 Inf. U. once on Day 57
  Arms: Group 2; Group 3
Biological: Placebo — One 0.5 ml IM injection of 0.9% saline administered once on Day 1 and Day 57
  Arms: Group 4

SUMMARY:
The purpose of this study is to demonstrate the non-inferiority of a heterologous prime-boost regimen using Ad26.ZEBOV as prime and MVA-BN-Filo as boost administered at different doses at a 56-day interval versus the same regimen with the recently released batches of Ad26.ZEBOV and MVA-BN-Filo in terms of humoral immune response against the Ebola virus (EBOV) GP (glycoprotein) as measured by enzyme-linked immunosorbent assay (ELISA) at 21 days post boost.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, parallel-group, multicenter study to evaluate safety and immunogenicity of Ad26.ZEBOV and MVA-BN-Filo at different dose levels, administered to healthy adults participants. The study consists of a Screening period of up to 6 weeks, vaccinations on Day 1 and Day 57, and a post-vaccination phase until the 6 months post-boost visit (Day 237). The participants will be randomized at baseline (on Day 1) in a 2:2:2:1 ratio to Groups 1, 2, 3 and 4. Safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion criteria :

* Must be healthy in the Investigator's clinical judgment on the basis of medical history, physical examination, electrocardiogram (ECG) and vital signs performed at Screening
* Must be healthy on the basis of clinical laboratory tests performed at Screening
* Before randomization, a woman must be either of childbearing potential and practicing (or intending to practice) a highly effective method of birth control consistent with local regulations regarding the use of birth control methods for participants participating in clinical studies, beginning at least 28 days prior to vaccination OR not of childbearing potential: postmenopausal [greater than (>)] 45 years of age with amenorrhea for at least 2 years or any age with amenorrhea for at least 6 months, and a serum follicle stimulating hormone (FSH) level >40 international unit per milliliter (IU/L); permanently sterilized (for example, bilateral tubal occlusion [which includes tubal ligation procedures as consistent with local regulations], hysterectomy, bilateral salpingectomy, bilateral oophorectomy); or otherwise be incapable of pregnancy
* Woman of childbearing potential must have a negative serum [beta-human chorionic gonadotropin (beta-hCG)] at Screening and a negative urine beta-hCG pregnancy test immediately prior to each study vaccine administration
* Man who is sexually active with a woman of childbearing potential and has not had a vasectomy performed more than 1 year prior to Screening must be willing to use condoms for sexual intercourse beginning prior to enrollment, in addition to the birth control method used by the female partner

Exclusion criteria:

* Having received a candidate Ebola vaccine
* Diagnosed with Ebola virus disease, or prior exposure to Ebola virus, including travel to West Africa less than 1 month prior to Screening. West Africa includes but is not limited to the countries of Guinea, Liberia, Mali, and Sierra Leone
* Having received any experimental candidate adenovirus serotype 26 (vector: Ad26) or Modified Vaccinia Ankara (MVA)- based vaccine in the past
* Known allergy or history of anaphylaxis or other serious adverse reactions to vaccines or vaccine products (including any of the constituents of the study vaccines) including known allergy to egg, egg products and aminoglycosides
* Presence of acute illness or temperature greater than or equal to (>=) 38.0 (°C) centigrade on Day 1

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 525 (Actual)
Dates: Start 2015-09-21 (Actual); Primary Completion 2016-06-07 (Actual); Study Completion 2016-11-29 (Actual)

PRIMARY OUTCOMES:
Immune Responses to the Study Vaccine Regimens against Ebola virus (EBOV) Glycoprotein (GP) using EBOV GP protein Enzyme-linked Immunosorbent Assay (ELISA) | At 21 days post boost vaccination
  The humoral immune response will be assessed by enzyme-linked immunosorbent assay (ELISA) binding antibody

SECONDARY OUTCOMES:
Immune Responses to the Study Vaccine Regimens against Ebola virus (EBOV) Glycoprotein (GP) using EBOV GP protein Enzyme-linked Immunosorbent Assay (ELISA) | At Days 1, 29, 57 post prime dose and at days 42, and 180 post boost vaccination
  The humoral immune response will be assessed by enzyme-linked immunosorbent assay (ELISA) binding antibody
Number of Participants with Solicited Local and Systemic Adverse Events (AEs) | Up to 7 days after each vaccination
Number of Participants with Adverse Events (AEs) | Up to 42 days post boost vaccination
Number of Participants with Serious Adverse Events (SAEs) | Continuous throughout the duration of study (Up to Day 237)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Vaccines & Prevention B.V. Clinical Trial, Study Director — Janssen Vaccines & Prevention B.V.
Locations (6):
- United States (6):
  - Huntsville, Alabama
  - San Diego, California
  - Melbourne, Florida
  - Peoria, Illinois
  - Mishawaka, Indiana
  - Rockville, Maryland

REFERENCES:
- [Derived] Bockstal V, Gaddah A, Goldstein N, Shukarev G, Bart S, Luhn K, Robinson C, Anumendem D, Leyssen M, Douoguih M. Assessments of different batches and dose levels of a two-dose Ad26.ZEBOV and MVA-BN-Filo vaccine regimen. NPJ Vaccines. 2021 Dec 20;6(1):157. doi: 10.1038/s41541-021-00402-8. PMID 34930928